CLINICAL TRIAL: NCT04018794
Title: Development of a Mobile App for an Executive Functioning Intervention for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAS# A127552
Record Dates: First submitted 2019-07-09; First posted 2019-07-15 (Actual); Results first posted 2021-11-19 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Attention Deficit Hyperactivity Disorder Symptoms

STUDY DESIGN:
Intervention Model Description: One group with behavioral/organizational skills intervention augmented with digital health application
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Behavioral/organizational skills intervention plus mobile app (Experimental): Behavioral/organizational skills intervention plus mobile application (16, 20-30 minute sessions, twice/weekly for 8 weeks)
  Interventions: Device: Behavioral/organizational skills intervention augmented with digital health application

INTERVENTIONS:
Device: Behavioral/organizational skills intervention augmented with digital health application — Behavioral/organizational skills intervention with digital health application augmentation

SUMMARY:
This study develops an initial prototype of a mobile tool that will support clinician-directed behavioral/organizational skills treatment for adolescents with Attention Deficit Hyperactivity Disorder (ADHD) with input guided from key stakeholders.

DETAILED DESCRIPTION:
Attention-Deficit/Hyperactivity Disorder (ADHD) is one of the most common childhood mental health disorders, affecting 7-9% of children and adolescents, and leading to substantial impairment in adolescence. Despite evidence suggesting that behavioral interventions are efficacious, approximately 40-60% of adolescents receiving behavioral treatment show little to no improvement and skills are rarely generalized beyond treatment sessions. Lack of adolescent motivation and engagement, between-session skills use, reward saliency, and family involvement are key contributors to these limited effects. Mobile digital health (dHealth) strategies and gamification techniques, offer unique opportunities for overcoming the barriers of treatments specific to ADHD by using interactive tools to reinforce in-vivo skill practice, providing opportunities for immediate reinforcement, and motivating adolescents with digital rewards. The primary goal of this study is to develop and preliminarily test the integration of a digital health tool into organizational/behavioral skills treatment for adolescents with ADHD by improving executive functioning skills, providing in-vivo skills reinforcement, and monitoring adolescents' skill utilization. The proposed research will use an iterative stakeholder-centered design to develop, refine, and preliminarily test a novel digital health tool, applied as an adjunct to behavioral treatment for adolescents with ADHD (ages 11-15). This includes focus groups with key stakeholders and an open preliminary feasibility trial and usability testing. Data collected from focus groups will inform what content and features could be developed to overcome challenges to adolescent engagement and parent involvement. During the open trial (N=20) we will assess intervention feasibility, usability, and acceptability. During and after the clinical trial, we will collect continuous feedback from users on the usability and utility of the tool. At the end of this study we will complete debugging and programming to maximize usability before a future larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* 1) Youth ages of 11-14 years (6-8th grade) that are attending a participating school
* 2) referred by SMHP as a youth with apparent ADHD-related problems,
* 3) ≥6 symptoms (item score ≥2) of Inattention or Hyperactivity-Impulsivity on the pooled parent and teacher Vanderbilt ADHD Rating Scale
* 4) ≥3 on the Impairment Rating Scale by parent and teacher (cross-situational impairment)
* 5) Parent consent and adolescent assent must be provided; b)

Exclusion Criteria:

* 1) No presence of conditions that are incompatible with this study's treatment including: Parent or adolescent report of a prior diagnosis of either Autism Spectrum Disorder, Bipolar Disorder, a Dissociative Disorder, Severe visual or hearing impairment, severe language delay or intellectual impairment, or a Psychotic Disorder will be excluded. Rationale: Individuals with these disorders often have very dysregulated behavior and impairments that deviate from the focus of this study.
* 2) Adolescent is in all-day special education classes or if core classes not in regular education classrooms. Rationale: The vast majority of adolescent with ADHD are served in regular education classrooms and students in full-day self-contained classrooms often have different challenges than students in regular education.
* 3) Adolescent planning to change (start or stop) psychotropic medication. Note: Adolescents taking medication will be required to meet all entry criteria, including impairment criteria, thus indicating a need for the intervention. Adolescent taking medication for attention or behavior are eligible as long as their medication regimens are stable. Participating parents will also need to be able to read/speak English because all measures are in English, and the intervention will be conducted in English.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa R Dvorsky, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited from local schools and enrolled were assigned to a single-arm/group where they all evaluated the usability and feasibility of the ATOM intervention tool as designed. Ratings of usability and feasibility were collected before and after using the ATOM tool.
Pre-assignment Details: All participants were assigned to a single-arm/group where they all evaluated the usability and feasibility of the ATOM intervention tool as designed. None were excluded upon enrollment.
Period: Overall Study
Arm/Group | Behavioral/Organizational Skills Intervention Plus Mobile App
Started | 15 (N=15 students participants completed the open trial of usability/feasibility of the intervention and completed quantitative ratings of usability before and after using the program.)
Completed | 15 (N=15 students participants completed the open trial of usability/feasibility of the intervention and completed quantitative ratings of usability before and after using the program.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Behavioral/Organizational Skills Intervention Plus Mobile App
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: System Usability Scale
Description: 10-item technology-agnostic scale assessing technology product usability. The total SUS score ranges from 0 to 100, with higher scores indicating higher usability. SUS scores above 80 indicated good usability. The SUS has high internal consistency (α=.91) and high convergent validity with a separate rating of usability and user satisfaction (r=.8). The present study will assess system usability at post-treatment (month 3).
Time Frame: at month 3 (1-month post-intervention)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Behavioral/Organizational Skills Intervention Plus Mobile App
Number analyzed (Participants) | 15
score on a scale | 71 [40 to 100]

2. Primary Outcome: Post Stakeholder Feasibility and Usability Rating
Description: 8-item Stakeholder Feasibility and Usability Rating (SFUR) was used to assess stakeholders' perceptions of the overall feasibility and usability of the program. The SFUR score is a mean of all items and ranges from 1 to 5, with higher scores indicating higher feasibility and usability. This measure was developed for the present study. The present study will assess these feasibility ratings at post-treatment (month 3).
Time Frame: at month 3 (1-month post-intervention)
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Behavioral/Organizational Skills Intervention Plus Mobile App
Number analyzed (Participants) | 15
units on a scale | 4.3 [1 to 5]

3. Other Pre Specified Outcome: Services Use in Children and Adolescents - Parent Interview (SCA-PI)
Description: SCA-PI (Hoagwood et al., 2004) will assess medication and psychosocial treatment use and changes in use including any school (e.g., Daily Report Card) or community services during the study from baseline/pre-treatment (month 0) to post-intervention (3 months).
Time Frame: Change from Baseline (month 0) to Post-Intervention (3 months)
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Demographics/Background Form
Description: A background form will collect information sufficient to calculate Hollingshead Socioeconomic Index as well as family income, marital status, and child's developmental and psychiatric history. Teachers and SMHPs will also complete a brief demographic form to assess age, race, and experience.
Time Frame: Baseline (month 0)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events were assessed at the time of data collection for each participant and monitored by the study coordinator and study staff.
Arm/Group | Behavioral/Organizational Skills Intervention Plus Mobile App
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT04018794/Prot_SAP_ICF_000.pdf